CLINICAL TRIAL: NCT05073315
Title: A Multicenter, Randomized, Double-blind Study Evaluating the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of Multiple Switches Between Humira® (Adalimumab [US]) and ABP 501 Compared With Continued Use of Adalimumab in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Comparative Study Between ABP 501 and Humira® in Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200497; 2021-000542-18 (EudraCT Number)
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Plaque Psoriasis
Keywords: Adalimumab; Biosimilars; Tumor necrosis factor; Psoriasis Area and Severity Index
MeSH Terms: interventions — Adalimumab; ABP 501

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study is double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continued-use Group (Adalimumab) (Active Comparator): Randomized participants will receive continuous injection of adalimumab Q2W until last dose at Week 28.
  Interventions: Drug: Adalimumab
- Switching Group (Adalimumab - ABP 501) (Experimental): Participants will initially receive adalimumab until Week 10 during the lead-in period. Thereafter, starting from Week 12, participants will switch between ABP 501 and adalimumab Q2W with last dose of ABP 501 at Week 28.
  Interventions: Drug: Adalimumab; Drug: ABP 501

INTERVENTIONS:
Drug: Adalimumab — Participants will receive subcutaneous (SC) injection of adalimumab
  Other Names: Humira®
Drug: ABP 501 — Participants will receive SC injection of ABP 501
  Arms: Switching Group (Adalimumab - ABP 501)

SUMMARY:
Study to evaluate pharmacokinetics, efficacy, safety and immunogenicity of multiple switches between Humira® and ABP 501 (new high concentration formulation) compared with continued use of Humira® in participants with moderate to severe plaque psoriasis. This multi-center study is composed of two periods: A lead-in period of treatment with Humira® followed by a randomized two parallel arm period.

ELIGIBILITY:
Inclusion Criteria:

* Participants has moderate to severe plaque psoriasis (with or without psoriatic arthritis) for at least 6 months and has stable disease for at least 2 months
* Participants has a score of PASI ≥ 12, involvement of ≥ 10% body surface area (BSA) and static Physician's Global Assessment (sPGA) ≥ 3 at screening and at baseline
* Participant has no known history of latent or active tuberculosis

Exclusion Criteria:

* Participant has erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication induced psoriasis, or other skin conditions at the time of screening (eg, eczema) that would interfere with evaluations of the effect of investigational product of psoriasis
* Participant has an active infection or history of infections
* Participant has received biologic treatment for psoriasis within the previous month or 5 drug half-lives (whichever is longer) prior to enrollment
* Participant has received nonbiologic systemic psoriasis therapy within 4 weeks prior to enrollment
* Participant has received ultraviolet (UV) A phototherapy (with or without psoralen) or excimer laser within 4 weeks prior to enrollment, or UV B phototherapy within 2 weeks prior to enrollment
* Participant has received topical psoriasis treatment within 2 weeks prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (88):
- United States (35):
  - Total Skin and Beauty Dermatology Center PC, Birmingham, Alabama
  - Johnson Dermatology Clinic, Fort Smith, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Revival Research, Doral, Florida
  - Altus Research, Inc., Lake Worth, Florida
  - International Dermatology Research, Inc, Miami, Florida
  - Tory Sullivan MD PA, North Miami Beach, Florida
  - Marietta dermatology skin care, Marietta, Georgia
  - Georgia Skin and Cancer Clinic - Clinic, Savannah, Georgia
  - NorthShore University HealthSystem Dermatology, Skokie, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Lawrence J Green, MD, LLC, Rockville, Maryland
  - ALLCUTIS Research, LLC., Beverly, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - David Fivenson, MD, PLC, Ann Arbor, Michigan
  - Henry Ford Health System - New Center One, Detroit, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Vivida Dermatology, Las Vegas, Nevada
  - Skin Search of Rochester, Inc., Rochester, New York
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Wright State Physicians, Inc, Fairborn, Ohio
  - Dermatologists of Southwest Ohio, Mason, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - University of Pittsburgh Medical Center/Falk Medical Center, Pittsburgh, Pennsylvania
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Bellaire Dermatology Associates (BDA), Bellaire, Texas
  - Center for Clinical Studies, LTD.LLP, Houston, Texas
  - Austin Institute for Clinical Research - Dermatology, Houston, Texas
  - Cutis Wellness Dermatology & Dermapathology, PLLC, Laredo, Texas
  - Progressive Clinical Research [Texas], San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
- Canada (15):
  - Beacon Dermatology, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - CCA Medical Research, Ajax, Ontario
  - SimcoDerm Medical & Surgical Dermatology Center, Barrie, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - DermEffects, London, Ontario
  - DermEdge Research Inc., Mississauga, Ontario
  - North Bay Dermatology Centre Inc., North Bay, Ontario
  - The Centre for Clinical Trials Inc., Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Toronto Research Centre - Dermatology, Toronto, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario
  - Dre Angélique Gagné-Henley MD inc, Saint-Jérôme, Quebec
- Estonia (3):
  - North Estonia Medical Centre, Tallinn, Harju
  - Clinical Research Center, Tartu, Tartu
  - Tartu University Hospital, Tartu, Tartu
- Germany (7):
  - Derma-Study-Center-FN, Friedrichshafen, Baden-Wurttemberg
  - Klinische Forschung Gruppe Nord (KFGN), Schwerin, Mecklenburg-Vorpommern
  - Hautzentrum im Jahrhunderthaus, Bochum, North Rhine-Westphalia
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - UKSH Campus Kiel - ZeH (Dermatologie), Kiel, Schleswig-Holstein
  - Rothhaar Studien GmbH, Berlin
  - TFS Trial Form Support GmbH, Hamburg
- Latvia (5):
  - Health Centre 4 Ltd., Diagnostics Centre, Riga, Rga
  - Riga 1st hospital, Clinic of Dermatology and STD, Riga, Rga
  - J.Kisis LtD, Riga, Rga
  - Health and Aesthetics Ltd, Riga
  - Smite Aija doctor practice in dermatology, venereology, Talsi
- Poland (23):
  - High-Med Przychodnia Specjalistyczna, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka, Warsaw, Masovian Voivodeship
  - ClinicMed Daniluk, Nowak Sp. J., Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Care Clinic SP. Z O.O., Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Pratia MCM Krakow, Krakow
  - Centrum Nowoczesnych Terapii "Dobry Lekarz" Sp. z o.o., Krakow
  - NZOZ ALL-MED Centrum Medyczne, Lodz
  - Centrum Terapii Wspolczesnej, J.M. Jasnorzewska S.K.A., Lodz
  - Centrum Zdrowia i Urody Maxxmed, Lublin
  - ETG Lublin, Lublin
  - Agnieszka Miasik-Pogodzinska DrDerm Centrum Medyczne, Nowy Targ
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Solumed Centrum Medyczne, Poznan
  - Clinical Research Center Sp. z o.o., Medic-R Sp. K., Poznan
  - Poradnia Dermatologiczno-Wenerologiczna MEDIDERM NZOZ, Torun
  - RCMed Oddzia Warszawa, Warsaw
  - Carpe Diem Centrum Medycyny Estetycznej, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - Ginemedica Sp. z o.o. Sp.k, Wroclaw
  - WroMedica I. Bielicka, A. Strzalkowska s.c., Wroclaw
  - Centrum Medyczne Oporow, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 425 participants were enrolled in the study at 83 centers across 6 countries (Canada, Estonia, Germany, Latvia, Poland, and the US) between October 2021 and December 2022.
Pre-assignment Details: Participants were enrolled in Period 1 of the study (Lead-in Period) and received adalimumab (Humira®) subcutaneously (SC) during a 12-week period. Participants who responded to treatment during Period 1 (achieving PASI ≥ 50) were randomized in Period 2 to either the Continued-use Group or the Switching Group. Period 2 lasted 20 weeks from Week 12 to Week 32.
Groups:
- Period 1 (Lead-in Period): Participants with plaque psoriasis (Ps) received adalimumab 100 mg/mL SC from Week 1 to Week 12 for a total of 6 doses (Week 1/Day 1 [80 mg], Week 2/Day 8 [40 mg], Week 4, Week 6, Week 8, and Week 10 [40 mg]) during the Lead-in Period.
- Period 2 (Switching Group): Participants with Ps who responded to treatment, defined as achieving PASI ≥ 50 in Period 1, were randomised to the Switching Group from Week 12 to Week 32 in Period 2 of the study. Participants received ABP 501 Q2W (Week 12 and Week 14 [40 mg]), adalimumab Q2W (Week 16 and Week 18 [40 mg]), and ABP 501 Q2W again (Week 20, Week 22, Week 24, Week 26, Week 28 [40 mg]).
- Period 2 (Continued-use Group): Participants with Ps who responded to treatment achieving PASI ≥ 50 in Period 1, were randomised to the Continued-use Group from Week 12 to Week 32 in Period 2 of the study. Participants continued receiving adalimumab 40 mg Q2W.
Period: Period 1 (Lead-in Period)
Arm/Group | Period 1 (Lead-in Period) | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Started | 425 | 0 | 0
Completed | 380 | 0 | 0
Not Completed | 45 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Did not Meet PASI 50 at Week 12 | 23 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Period: Period 2
Arm/Group | Period 1 (Lead-in Period) | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Started | 0 | 186 | 194
Completed | 0 | 174 | 173
Not Completed | 0 | 12 | 21
Not completed — Adverse Event | 0 | 3 | 6
Not completed — Lost to Follow-up | 0 | 5 | 5
Not completed — Withdrawal by Subject | 0 | 4 | 9
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data is reported for the Safety Analysis Set and reflects data collected at baseline for the switching and continued use groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group) | Total
Number analyzed (Participants) | 186 | 194 | 380
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (13.27) | 44.3 (13.91) | 44.6 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 63 | 119
  Male | 130 | 131 | 261
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 36 | 63
  Not Hispanic or Latino | 158 | 158 | 316
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 14 | 10 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 162 | 172 | 334
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 Over the Dosing Interval (AUCtau) of ABP 501 (Switching Group) and Adalimumab (Continued-use Group)
Description: Participants analyzed according to actual treatment received.
Time Frame: Week 28 pre-dose and 1hour, 1 day, 3 days, 4 days, 7 days, 11 days, and 14 days post Week 28 dose
Population: The Pharmacokinetic (PK) Parameter Analysis Set consists of all randomized participants who receive at least one dose post-randomization and who have an evaluable ABP 501 or adalimumab serum concentration-time profile between Weeks 28 and 30.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 146 | 145
hr*μg/mL | 1458.03 (156.6) | 1472.68 (174.9)
Statistical Analysis 1: Comparison: Period 2 (Switching Group) vs Period 2 (Continued-use Group); Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Ratio Geometric Least Square Mean (GMR) = 1.0516, 90% CI 2-sided [0.9010 to 1.2273]

2. Primary Outcome: Maximum Serum Concentration (Cmax) of ABP 501 (Switching Group) and Adalimumab (Continued-use Group)
Description: Participants analyzed according to treatment received.
Time Frame: Week 28 pre-dose, 1h post Week 28 dose, 1 day post Week 28 dose, 3 days, 4 days, 7 days, 11 days, and 14 days post Week 28 dose
Population: The PK Parameter Analysis Set consists of all randomized participants who receive at least one dose post-randomization and who have an evaluable ABP 501 or adalimumab serum concentration-time profile between weeks 28 and 30.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 153 | 153
μg/mL | 4.91 (153.6) | 5.01 (160.4)
Statistical Analysis 1: Comparison: Period 2 (Switching Group) vs Period 2 (Continued-use Group); Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Least Square Mean Ratio = 1.0044, 90% CI 2-sided [0.8717 to 1.1574]

3. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of ABP 501 (Switching Group) and Adalimumab (Continued-use Group)
Description: Time to reach maximum serum concentration.
Time Frame: as for outcome 2
Population: The analyses of the secondary PK endpoints is based on the PK Concentration Analysis Set, which included all randomized participants who received at least 1 dose of investigational product (IP) post-randomization and had at least 1 reported serum concentration of ABP 501 or adalimumab on or after the day of randomization.
Measure: Median (Full Range); unit: Hours
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 162 | 160
Hours | 72.30 [0 to 266.5] | 72.35 [0 to 334.9]

4. Secondary Outcome: Trough Concentration (Ctrough) of ABP 501 (Switching Group) and Adalimumab (Continued-use Group)
Time Frame: Pre-dose at Week 12, Week 16, Week 20, and Week 28
Population: The analyses of the secondary PK endpoints is based on the PK Concentration Analysis Set, which included all randomized participants who received at least 1 dose of IP post-randomization and had at least 1 reported serum concentration of ABP 501 or adalimumab on or after the day of randomization. All participants reported in the overall number of participants analyzed contributed data to this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 162 | 160
ng/mL
  Week 12: number analyzed (Participants) | 153 | 153
  Week 12 | 4528.7316 (88.9) | 4072.5556 (119.0)
  Week 16: number analyzed (Participants) | 150 | 151
  Week 16 | 4046.3069 (144.1) | 3682.0016 (188.1)
  Week 20: number analyzed (Participants) | 143 | 141
  Week 20 | 4113.0839 (160.8) | 4332.1272 (148.9)
  Week 28: number analyzed (Participants) | 140 | 135
  Week 28 | 3736.9917 (182.1) | 4014.4980 (193.5)

5. Secondary Outcome: PASI Percent Improvement From Baseline (Day 1) to Week 30
Description: The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
  Percent improvement from baseline was calculated as (value at baseline - value at post-baseline visit) × 100 / (value at baseline).
Time Frame: Baseline (Day 1) and Week 30
Population: Based on the per-protocol (PP) efficacy analysis set as observed, which consisted of all participants who were randomized and received all assigned doses post randomization and who had not experienced an important protocol deviation that could affect the efficacy endpoints; used for primary analysis of the secondary efficacy endpoints; analyzed according to actual treatment received.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 151 | 151
Percentage Change | 88.56 [86.07 to 91.05] | 91.01 [88.76 to 93.26]
Statistical Analysis 1: Comparison: Period 2 (Switching Group) vs Period 2 (Continued-use Group); Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Mean Difference (Final Values) = -2.47, 90% CI 2-sided [-5.23 to 0.29]

6. Secondary Outcome: Number of Participants Achieving PASI 75 Response at Week 30
Description: A PASI 75 response is a 75% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline (Day 1) and Week 30
Population: Based on the PP efficacy analysis set, which consisted of all participants who were randomized and received all assigned doses post randomization and who had not experienced an important protocol deviation that could affect the efficacy endpoints; used for primary analysis of the secondary efficacy endpoints; analyzed according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 151 | 151
Participants | 131 | 134

7. Secondary Outcome: Number of Participants Achieving PASI 90 Response at Week 30
Description: A PASI 90 response is a 90% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline (Day 1) and Week 30
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 151 | 151
Participants | 92 | 108

8. Secondary Outcome: Number of Participants Achieving PASI 100 Response at Week 30
Description: A PASI 100 response is a 100% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline (Day 1) and Week 30
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 151 | 151
Participants | 52 | 61

9. Secondary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAE)
Description: TEAEs are any event that occurred after the participant received study treatment. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration were recorded as TEAEs.
  A serious TEAE is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment(s) that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Time Frame: Baseline up to Week 32
Population: Population from the Safety Analysis Set (SAS). Population consisted of participants who were randomized and received at least 1 dose of IP post randomization; used for analyses of the safety endpoints during the Post-randomization Period; analyzed according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 186 | 194
Participants
  TEAE | 97 | 106
  Serious TEAE | 3 | 4

10. Secondary Outcome: Number of Participants Experiencing Events of Interest (EOI)
Description: An EOI is defined as a noteworthy event for a particular product or class of products that a sponsor may wish to monitor carefully. It could be serious or non-serious and could include events that might be potential precursors or prodromes for more serious medical conditions in susceptible individuals.
Time Frame: Baseline up to Week 32
Population: Population from the SAS. Population consisted of participants who were randomized and received at least 1 dose of IP post randomization; used for analyses of the safety endpoints during the Post-randomization Period; analyzed according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 186 | 194
Participants | 13 | 17

11. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Expression Post Randomization
Description: Anti-drug antibody samples were drawn prior to investigational product administration at dosing visits.
Time Frame: Week 16, Week 20, Week 28, Week 30, and Week 32
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2 (Switching Group) | Period 2 (Continued-use Group)
Number analyzed (Participants) | 186 | 194
Participants
  Participants with a post-randomization result | 186 | 194
  Binding antibody negative or no result prior to the first dose of post-randomization IP | 25 | 18
  Binding antibody positive with negative/no result prior to first dose post-randomization | 16 | 10
  Transient binding antibody positive with negative/no result prior to first dose post-randomization | 3 | 2
  Neutralizing antibody negative or no result prior to the first dose of post-randomization IP | 174 | 182
  Neutralizing antibody positive with negative/no result prior to first dose post-randomization | 21 | 27
  Transient neutralizing antibody positive with negative/no result prior first dose post-randomization | 2 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to 32 weeks
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Period 1 (Lead-in Period): Participants with Ps received adalimumab 100 mg/mL SC from Week 1 to Week 12 for a total of 6 doses (Week 1/Day 1 [80 mg], Week 2/Day 8 [40 mg], Week 4, Week 6, Week 8, and Week 10 [40 mg]) during the Lead-in Period.
Arm/Group | Period 1 (Lead-in Period) | Period 2 (Continued-use Group) | Period 2 (Switching Group)
All-Cause Mortality (participants affected / at risk) | 1/425 | 0/194 | 0/186
Serious Adverse Events (participants affected / at risk) | 5/425 | 4/194 | 3/186
Other Adverse Events (participants affected / at risk) | 38/425 | 28/194 | 26/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 (Lead-in Period) (N=425) | Period 2 (Continued-use Group) (N=194) | Period 2 (Switching Group) (N=186)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Trigeminal nerve disorder (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 (Lead-in Period) (N=425) | Period 2 (Continued-use Group) (N=194) | Period 2 (Switching Group) (N=186)
COVID-19 (Infections and infestations) | 14 | 7 | 13
Nasopharyngitis (Infections and infestations) | 12 | 11 | 13
Headache (Nervous system disorders) | 16 | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT05073315/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT05073315/SAP_002.pdf